CLINICAL TRIAL: NCT06810947
Title: Evaluation of Treatments for Allergic Rhinitis
Brief Title: Evaluation of Treatments for Allergic Rhinitis (Rhinal 2)
Acronym: RHINAL 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Vitrobio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2024 PICKERING
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-12

CONDITIONS: Allergic Rhinitis
Keywords: post-market; clinical study; follow up; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: 2 indépendants parallel groups (Product A and B) treating a common pathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment using medical device A (Experimental): Treatment using medical device A (ALLERSPRAY G), it's a topically applied liquid filmogen bandage (in the form of a hypertonic slightly viscous liquid solution) for the treatment of ALLERGIC RHINITIS OF VARIOUS ORIGINS.
  Interventions: Device: ALLERSPRAY-G (device A)
- Treatment using medical device B (Experimental): Treatment using medical device B (PCNS), it's a topically applied liquid filmogen bandage (in the form of a hypertonic slightly viscous liquid solution) for the treatment of ALLERGIC RHINITIS OF VARIOUS ORIGINS.
  Interventions: Device: PCNS (device B)

INTERVENTIONS:
Device: ALLERSPRAY-G (device A) — Symptomatic treatment consists of 3 sprays of medical device A in each nostril while breathing in slightly. This process should be repeated 4 times a day for 14 days by patients participating in the study.
  Arms: Treatment using medical device A
Device: PCNS (device B) — Symptomatic treatment consists of 3 sprays of medical device B in each nostril while breathing in slightly. This process should be repeated 4 times a day for 14 days by patients participating in the study.
  Arms: Treatment using medical device B

SUMMARY:
The goal of this clinical study is to perform a post-market clinical follow-up of 2 medical devices (liquid bandage in the form of a spray : ALLERSPRAY G (product A - code AAG), PCNS (product B - code PC) indicated for symptomatic treatment of allergic rhinitis. This follow-up will consist in collecting real-life clinical data to confirm the safety and efficacy of medical devices used in the treatment of allergic rhinitis of adults patients while allowing an assessment of the product's risk/benefit ratio.

The main questions it aims to answer are:

* Primary objective : Evaluate in real life the tolerance of medical device A and B used in the treatment of allergic rhinitis.
* Secondary objectives : Evaluate the efficacy of medical device A and B on allergic rhinitis and the quality of life using the device A and B.

No comparison group will be constituated because of the type of study (post market follow up) and no comparison between device A and B will be done.

58 participants (29 for medical device A and 29 for medical device B) with allergic rhinitis will be asked to :

* use medical device A or B during 2 weeks (from inclusion visit to end of study visit),
* complete each day at home a diary (recording intensity of 4 nasal symptoms, adverse events, concomitant treatments),
* complete " Quality of life evaluation (sleep, daily activities, fatigue, irritability) " at inclusion visit and end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* " Score For Allergic Rhinitis " ≥ 8
* Age ≥ 18
* Able to refrain from using any treatment for allergic rhinitis or any other treatment that could interfere with the purpose of the study,
* Effective contraception for women of reproductive age,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance to give written consent and inscription to VRB french platform for the duration of the study,
* Affiliation to the French Social Security system,

Exclusion Criteria:

* Known hypersensitivity to any of the components of the evaluated products,
* Use of any treatment to treat allergic rhinitis,
* pregnant or breastfeeding women,
* participating in another clinical trial, or being in the exclusion period, or having received a total amount of benefits exceeding EUR 6000 over the 12 months preceding the start of the trial,
* benefiting from a measure of legal protection (guardianship, deprivation of liberty, safeguard of justice),
* having a medical and / or surgical history judged by the investigator or his representative to be incompatible with the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | From visit 1 (day 1) to the end of treatment at day 14
  Recording of all adverse events on an electronic journal

SECONDARY OUTCOMES:
Total nasal symptom score (TNSS) | basal and twice a day from visit 1 (day 1) to the end of treatment at day 14
  4 symptoms (stuffy nose, runny nose, sneezing, itching nose) will be evaluated (from 0 "no embarassement" to 10 "extremely embarrassed") by the patient every day during the treatment period (from day 1 to day 14). the 4 symptoms composed the total nasal symptom score (TNSS). Basal and the mean last 3 days of treatment TNSS score of will be compared.
Impact of allergic rhinitis on sleep | basal (day 1) and after the study treatment period (day 15)
  Evaluation of how much your allergic rhinitis and associated symptoms interfere/impact on sleep (from 0 (not annoying/not at all impact) and 10 (extremely annoying/very impacted) on a visual analog scale
Impact of allergic rhinitis on daily activities | basal (day 1) and after the study treatment period (day 15)
  Evaluation of how much your allergic rhinitis and associated symptoms interfere/impact on daily activities (from 0 (not annoying/not at all impact) and 10 (extremely annoying/very impacted) on a visual analog scale
Impact of allergic rhinitis on fatigue | basal (day 1) and after the study treatment period (day 15)
  Evaluation of how much your allergic rhinitis and associated symptoms interfere/impact on fatigue (from 0 (not annoying/not at all impact) and 10 (extremely annoying/very impacted) on a visual analog scale
Impact of allergic rhinitis on irritability | basal (day 1) and after the study treatment period (day 15)
  Evaluation of how much your allergic rhinitis and associated symptoms interfere/impact on irritability (from 0 (not annoying/not at all impact) and 10 (extremely annoying/very impacted) on a visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France